CLINICAL TRIAL: NCT00669929
Title: Cost-Effectiveness Analysis of Rotavirus Vaccination for Children in Korea
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Severance Hospital (Other)
Responsible Party: Yonsei University Health System Severance Hospital, Yonsei University
Other Study IDs: rota-001; yonsei-rota
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Gastroenteritis; Rotavirus Vaccines; Cost-Effectiveness
Keywords: Cost effectiveness analysis of rotavirus vaccination
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: patients visited to Severance hospital
- 2: patients visited to Youngdong Severance hospital
- 3: patients visited to Wonju Christian hospital

SUMMARY:
The primary objective of the proposed project is to estimate the economic impact of a national rotavirus immunization program in preventing rotavirus diarrhea among Korean children.

DETAILED DESCRIPTION:
Rotavirus is the leading cause of severe acute diarrhea or gastroenteritis among young children worldwide. In the first 5 years of life, about 90% of children experience at least one episode of rotavirus infection.Each year, rotavirus diarrhea is responsible for 440,000 deaths, 2 million hospitalizations, and 25 million outpatient visits among children younger than 5 years worldwide. In South Korea, rotavirus diarrhea rarely causes mortality, but it cause significant morbidity. A recent population-based study in Korea has estimated that the annual incidence of rotavirus diarrhea accounts for 56.9 cases per 1,000 children less than 5 years old. Oral, live pentavalent human-bovine reassortant rotavirus vaccine has been developed and licensed for the use of preventing rotavirus disease in many countries. Yet, there has been no research done to assess the impact of national rotavirus immunization program in Korea. It is expected that systematic appraisal on the national burden of rotavirus infection and potential public health and economic benefits of rotavirus vaccination for children in Korea will assists health policy makers to set a priority for the prevention of this disease.

ELIGIBILITY:
Inclusion Criteria:

* children aged under 5 years and diagnosed as acute gastroenteritis

Exclusion Criteria:

* none

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients to visit assigned hospital
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-06 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
patients' cost | one year

CONTACTS AND LOCATIONS:
Overall Officials: Dong Soo Kim, MD, PhD, Principal Investigator — professor
Locations (3):
- South Korea (3):
  - Wonju Christian Hospital, Wŏnju, Gangwon-do
  - Yonsei University Health System Severance Hospital, Seoul
  - Youngdong Severance Hospital, Seoul

REFERENCES:
- [Background] Hong SK, Lee SG, Lee SA, Kang JH, Lee JH, Kim JH, Kim DS, Kim HM, Jang YT, Ma SH, Kim SY, Paik SY. Characterization of a G11,P[4] strain of human rotavirus isolated in South Korea. J Clin Microbiol. 2007 Nov;45(11):3759-61. doi: 10.1128/JCM.01505-07. Epub 2007 Aug 29. PMID 17728473
- [Background] Kim DS, Lee TJ, Kang JH, Kim JH, Lee JH, Ma SH, Kim SY, Kim HM, Shin SM. Immunogenicity and safety of a pentavalent human-bovine (WC3) reassortant rotavirus vaccine in healthy infants in Korea. Pediatr Infect Dis J. 2008 Feb;27(2):177-8. doi: 10.1097/INF.0b013e31815aba79. PMID 18174862
- [Background] Lu CY, Lauderdale TL, Fang YH, Wang CY, Ho YH, Hung CL, Chang LY, Lee CY, Huang LM. Disease burden and related medical costs of rotavirus infections in Taiwan. BMC Infect Dis. 2006 Dec 15;6:176. doi: 10.1186/1471-2334-6-176. PMID 17173677